CLINICAL TRIAL: NCT05959291
Title: Free-HER: Discontinuation of Maintenance HER-2 Directed Therapy in Long-Term Survivors of Metastatic HER-2 Positive Breast Cancer
Brief Title: Discontinuation of Maintenance HER-2 Directed Therapy in Long-Term Survivors of Metastatic HER-2 Positive Breast Cancer
Acronym: Free-HER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Elisa Krill Jackson, Staff Physician, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20221166
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Metastatic Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-HER-2 Group (Experimental): Participants in this group will be monitored to see if patients discontinuing maintenance of anti-HER-2 treatments with ctDNA monitoring in addition to radiologic imaging and routine blood work will stay in complete radiological remission. Participants will be in this group for up to 3 years.
  Interventions: Other: Discontinuation of Anti-HER-2 Maintenance Treatment

INTERVENTIONS:
Other: Discontinuation of Anti-HER-2 Maintenance Treatment — Patients assigned to this group will be asked to discontinue anti-HER-2 maintenance treatment.

SUMMARY:
The purpose of this preliminary research study is to see if patients discontinuing maintenance Herceptin and/or other anti-HER-2 treatments with monitoring in addition to radiologic imaging and routine blood work will stay in complete radiological remission and to determine how long patients are able to stay in complete radiological remission without treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of HER-2 positive metastatic (Stage IV) breast cancer.
2. Patients in complete radiological remission (CRR), including a stable bone scan, as determined by computed tomography (CT), positron-emission tomography (PET), or PET-CT.

   a. Patients with brain metastasis are allowed to participate as long as their disease has been treated and radiologically stable for at least 36 months.
3. Patients must be on the same or current anti-HER-2 directed therapy for at least 36 months.
4. Archived tumor biopsy available.
5. Patients with no evidence of circulating tumor deoxyribonucleic acid (ctDNA) as determined by the Signatera assay.
6. Patients willing to stop maintenance anti-HER-2 directed therapy with close monitoring.
7. Patients with an Eastern Cooperative Oncology Group (ECOG) performance score from 0 to 2.
8. Patients ≥ 18 years of age.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with uncontrolled metastatic disease.
2. Patients whose disease has been controlled for less than 36 months on the same or current anti-HER-2 therapy.
3. Patients who are currently receiving or have received treatment for a secondary cancer other than resected non-melanoma skin cancer lesions or in situ cancer within the past 24 months.
4. Patients positive for ctDNA (which occurs when a patient's blood sample contains ≥2 target markers) with the Signatera assay.
5. Use of investigational drugs ≤ 28 days prior to study enrollment and during the study.
6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or that makes participation in the trial to be not in the best interest of the patient in the opinion of the Investigator.
7. Patients with impaired decision-making capacity.

Patients who are found to be ctDNA+ at study entry will be recorded as a screen failure (Section 5.4). Their Signatera testing results will be provided to their treating physician to aid in clinical decision-making for disease management and treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of maintaining remission after discontinuing use of anti-HER-2 | Up to 72 months
  The feasibility of maintaining remission of HER-2 will be measured as the proportion of patients who discontinue anti-HER-2 therapy and who remain in remission is assessed by monitoring ctDNA in the blood.

SECONDARY OUTCOMES:
Ability of re-attain remission after ctDNA+ status | Up to 72 months
  Ability to re-attain remission after ctDNA+ status is defined as returning to ctDNA- status within 6 months after testing ctDNA+ during the study. This is assessed by the monitoring of ctDNA in the blood of participants that have tested ctDNA positive after stopping anti-HER-2 maintenance therapy and chose to restart anti-HER-2 therapy.
Duration of response (DOR) | Up to 72 months
  The duration of response (DOR) in study participants that have restarted anti-HER-2 therapy measures the time from is ctDNA+ status to overall response rate (ORR). This includes study participants that have ctDNA+ status and have chosen to either restart their previous anti-HER-2 maintenance therapy or have started a new anti-HER-2 therapy. The ORR is determined by blood and imaging monitoring.
Diagnostic Accuracy of ctDNA Monitoring Assay to Identify Disease Progression | Up to 72 months
  Diagnostic accuracy is evaluated by comparing disease relapse and/or progression confirmed by imaging compared to study participants ctDNA status.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Krill Jackson, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No